CLINICAL TRIAL: NCT06064487
Title: Role of Renal Cell Arrest and Damage Biomarkers in Progression and Outcome of Sepsis Associated AKI
Brief Title: Renal Cell Arrest and Damage Biomarkers in Progression and Outcome of Septic AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: markers of septic AKI
Record Dates: First submitted 2023-09-21; First posted 2023-10-03 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: AKI - Acute Kidney Injury
Keywords: AKI; sepsis; markers; urine sediment
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Intervention Model Description: The current study will include 80 patients with sepsis associated AKI stage
  1 or 2 according to KDIGO definition admitted to Alexandria Main University Hospital. Urinary TIMP2 and IGFBP7: will be measured by the ELISA technique. Urinary KIM-1: will be measured by the ELISA technique. Examination of urine sediment from fresh urine sample.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- septic AKI patients (Experimental): 80 patients with sepsis associated AKI stage 1 or 2 according to KDIGO definition
  Interventions: Diagnostic Test: renal cell arrest and damage biomarkers assessment

INTERVENTIONS:
Diagnostic Test: renal cell arrest and damage biomarkers assessment — measurement of TIMP2 and IGFBP7, KIM-1

SUMMARY:
The aim of the current study is to assess the predictive value of renal cell arrest biomarkers (urinary TIMP2 and IGFBP7), renal damage biomarkers (urinary KIM-1) and microscopic examination of urinary sediment in progression and outcome of sepsis associated AKI.

DETAILED DESCRIPTION:
Acute kidney injury occurred in about 45-53% of patients with sepsis, and most septic AKI was mild or moderate AKI (KDIGO stage 1 or stage 2).

However, previous study showed that up to 40% of these mild or moderate AKI would progress to more severe AKI (KDIGO stage 3), of which 30% required dialysis and the risk of death increased by 3-fold, as high as 70%. Therefore, early identifying patients at high risk for progressive AKI might help clinicians to enhance individualized monitoring and personalized management in patient with septic AKI, which might prevent or halt the ongoing renal injury and improve the outcome of patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* AKI stage 1 or 2 according to KDIGO definition.
* Sepsis is defined based on the third international consensus definitions for sepsis and septic shock (Sepsis-3) as life threatening organ dysfunction caused by a dysregulated host response to infection. At least two of systemic inflammatory response syndrome (SIRS) criteria should be present

Exclusion Criteria:

* Age less than 18 years.
* Patients with pre-existing chronic kidney disease (eGFR<60 ml/min/1.73m2).
* Previous renal replacement therapy.
* Acute kidney injury caused by permanent postrenal obstruction.
* Pregnancy.
* Hepatorenal syndrome.
* Renal transplant recipients.
* Patients for whom survival to 30 days is unlikely due to end stage disease (end stage liver or heart disease or untreatable malignancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Urinary TIMP2 and IGFBP7 estimation | 90 days
  both will be measured by the ELISA technique
Urinary KIM-1 estimation | 90 days
  will be measured by the ELISA technique
Examination of urine sediment | 7 days
  by calculating Perazella score
progression of AKI | 90 days
  by assessing change in eGFR
Examination of urine sediment | 7 days
  by calculating Chawla score

SECONDARY OUTCOMES:
need for renal replacement therapy | 90 days
  need of any dialysis modality
mortality | 90 days
  death
length of ICU and hospital stay | 90 days
  duration of stay

CONTACTS AND LOCATIONS:
Overall Officials: Hala S ElWakil, MD, Study Chair — professor; salah s naga, MD, Principal Investigator — professor; Mohamed mamdouh Elsayed, MD, Study Chair — Lecturer; Mona m tahoun, MD, Study Chair — Lecturer; ahmed E El-deeb, Master, Study Chair — assistant lecturer
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Background] Maizel J, Daubin D, Vong LV, Titeca-Beauport D, Wetzstein M, Kontar L, Slama M, Klouche K, Vinsonneau C. Urinary TIMP2 and IGFBP7 Identifies High Risk Patients of Short-Term Progression from Mild and Moderate to Severe Acute Kidney Injury during Septic Shock: A Prospective Cohort Study. Dis Markers. 2019 Apr 1;2019:3471215. doi: 10.1155/2019/3471215. eCollection 2019. PMID 31061681
- [Background] Gunnerson KJ, Shaw AD, Chawla LS, Bihorac A, Al-Khafaji A, Kashani K, Lissauer M, Shi J, Walker MG, Kellum JA; Sapphire Topaz investigators. TIMP2*IGFBP7 biomarker panel accurately predicts acute kidney injury in high-risk surgical patients. J Trauma Acute Care Surg. 2016 Feb;80(2):243-9. doi: 10.1097/TA.0000000000000912. PMID 26816218
- [Derived] Elsayed MM, Eldeeb AE, Tahoun MM, El-Wakil HS, Naga SS. Does combining urine sediment examination to renal cell arrest and damage biomarkers improve prediction of progression and mortality of sepsis associated acute kidney injury? BMC Nephrol. 2025 Apr 17;26(1):195. doi: 10.1186/s12882-025-04096-1. PMID 40247231